CLINICAL TRIAL: NCT02594176
Title: A Randomised, Double-blind, Placebo Controlled Study of Topical FLEXISEQ® for the Treatment of Osteoarthritis of the Knee in Patients Contraindicated for or With Clinical Intolerance to NSAIDs
Brief Title: Study of FLEXISEQ® for Treatment of Osteoarthritis of the Knee in NSAID-compromised Patients
Acronym: OANIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pro Bono Bio (Industry)
Collaborators: International Medical Research - Partner GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-064-IV-01 (IMR-062)
Record Dates: First submitted 2015-10-20; First posted 2015-11-02 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Pain; NSAID; Sequessome
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): 2.2 g FLEXISEQ® twice daily
  Interventions: Device: FLEXISEQ®
- Placebo (Placebo Comparator): 2.2 g placebo twice daily
  Interventions: Device: Placebo

INTERVENTIONS:
Device: FLEXISEQ® — applicable gel
  Arms: Test Product
Device: Placebo — applicable gel
  Arms: Placebo

SUMMARY:
Primary Objective To substantiate the efficacy of 2.2 g FLEXISEQ® for the treatment of pain related to osteoarthritis (OA) of the knee in patients contraindicated for or with clinical intolerance to NSAIDs.

Secondary Objectives

* To substantiate the efficacy of 2.2 g FLEXISEQ® for the treatment of stiffness and improvement of joint function in patients contraindicated for or with clinical intolerance to NSAIDs and with OA of the knee.
* To substantiate safety and tolerability of 2.2 g FLEXISEQ® in patients contraindicated for or with clinical intolerance to NSAIDs and with OA of the knee.

DETAILED DESCRIPTION:
This post marketing clinical follow-up, randomised, double-blind study comparing the efficacy and tolerability of topical FLEXISEQ® with placebo for the treatment of osteoarthritis of the knee in patients contraindicated for or with clinical intolerance to NSAIDs and with OA of the knee will have a total individual treatment period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-mandated procedure
2. Willing and able to comply with study requirements
3. Outpatients with an age ≥ 50 (starting from the day after the 50th birthday)
4. Patient for whom their knee pain is the worst pain in the body and is able to identify the predominantly painful (target) knee
5. Patient has a primary diagnosis of Functional Class I-III OA of the target knee and patient meets American College of Rheumatology (ACR) clinical classification criteria for osteoarthritis of the knee
6. NSAID contraindicated or clinically intolerant
7. Females able to conceive (including peri-menopausal women who have had a menstrual period within 1 year) must be using appropriate birth control (defined as a method which results in a low failure rate
8. If female and able to conceive, patient has a negative urine pregnancy test at screening

Exclusion Criteria:

* General exclusion criteria

  1. Planned treatment or treatment with another investigational drug within 30 days prior to randomisation
  2. Patients who are inmates of psychiatric wards, prisons, or other state institutions
  3. Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
  4. Pregnancy or lactation
  5. Any planned or expected hospitalisation within the study period
  6. Patients not able to perform the WOMAC test (physically handicapped or immobile patient, e.g. wheel-chair bound)
  7. Any health condition which, in the investigator's opinion means the patient is likely to be unable to complete the 12 week study Medical history related exclusion criteria
  8. Skin lesions or dermatological diseases in the treatment area
  9. Extreme obesity (BMI > 35)
  10. Uncontrolled hypertension
  11. Requiring dialysis
  12. Hepatocellular insufficiency preventing use of paracetamol
  13. Alcohol abuse
  14. Intolerance to paracetamol
  15. Malignancy within the past 2 years
  16. Morbus Meulengracht/Gilbert Syndrome
  17. Neurological or psychiatric disorders compromising pain rating by the patient, such as but not limited to depressive disorders, schizophrenia or epilepsy
  18. Any other pain condition requiring acute or chronic use of pain medication that cannot be discontinued at screening
  19. Inflammatory arthritis including rheumatoid arthritis, psoriatic arthritis, gout, pseudo gout, systemic lupus erythematodes, ankylosing spondylitis, mixed connective tissue disease
  20. Symptomatic hip OA ipsilateral to the target knee
  21. Severe (axial misalignment > 10°), uncorrected genu vara and genu valga
  22. Arthroscopy of the target knee within 6 months prior or during the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
WOMAC pain score | 3 months
  Change from baseline to final visit of the average of the WOMAC pain subscale scores

SECONDARY OUTCOMES:
Patient Global Assessment of Change (PGIC) | 3 months
  PGIC-Score at final visit
WOMAC function score | 3 months
  Change from baseline to final visit of the average of the WOMAC function subscale scores
WOMAC stiffness score | 3 months
  Change from baseline to final visit of the average of the WOMAC stiffness subscale scores

OTHER OUTCOMES:
Adverse Events (AE) | 3 months
  Frequency of treatment emergent AEs per treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Rother, MD, Study Director — International Medical Research - Partner GmbH
Locations (1):
- IMR-Site #1-30, Gräfelfing, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conaghan PG, Dickson J, Bolten W, Cevc G, Rother M. A multicentre, randomized, placebo- and active-controlled trial comparing the efficacy and safety of topical ketoprofen in Transfersome gel (IDEA-033) with ketoprofen-free vehicle (TDT 064) and oral celecoxib for knee pain associated with osteoarthritis. Rheumatology (Oxford). 2013 Jul;52(7):1303-12. doi: 10.1093/rheumatology/ket133. Epub 2013 Mar 28. PMID 23542612
- [Background] Rother M, Conaghan PG. A randomized, double-blind, phase III trial in moderate osteoarthritis knee pain comparing topical ketoprofen gel with ketoprofen-free gel. J Rheumatol. 2013 Oct;40(10):1742-8. doi: 10.3899/jrheum.130192. Epub 2013 Sep 1. PMID 23996292
- [Background] Kneer W, Rother M, Mazgareanu S, Seidel EJ; European IDEA-033 study group. A 12-week randomized study of topical therapy with three dosages of ketoprofen in Transfersome(R) gel (IDEA-033) compared with the ketoprofen-free vehicle (TDT 064), in patients with osteoarthritis of the knee. J Pain Res. 2013 Oct 25;6:743-53. doi: 10.2147/JPR.S51054. eCollection 2013. PMID 24187510